CLINICAL TRIAL: NCT00165425
Title: Cardiac Screening in Survivors of Hodgkin's Disease Treated With Mediastinal Irradiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrea K. Ng, MD, Professor of Radiation Oncology, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-295
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hodgkin's Disease
Keywords: Cardiac screening; Cardiac stress test; Echocardiogram
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac screening (Experimental): Interventions:
  Participants will
  * meet with study cardiologist
  * undergo cardiac risk factors screening
  * undergo resting and stress echocardiogram (echo and stress echo)
  Interventions: Procedure: Echo/Stress Echo

INTERVENTIONS:
Procedure: Echo/Stress Echo — Participants will under resting echocardiogram and stress echocardiogram (echo and stress echo) and the results will be interpreted by a cardiologist

SUMMARY:
The main purpose of this study is to determine if it is possible to put into practice a cardiac screening program for survivors of Hodgkin's disease. In this study, we would also like to screen for cardiac risk factors that can be modified either through life-style changes or medications, to uncover significant abnormal heart findings in which treatments may be needed, and to see if there is a link between cardiac health and quality of life.

DETAILED DESCRIPTION:
* On the day of the patient's scheduled follow-up visit with their oncologist, additional blood work will be obtained and the patient will fill out questionnaires concerning their general health and assessing quality of life.
* A separate cardiology visit with a preventative cardiologist will be performed. At this visit, the patient will undergo a Stress Echocardiogram.
* A Stress Echocardiogram is made up of three parts: Resting echo study, stress test and repeat echo while the heart is still beating fast.
* A resting echo provides the baseline examination and demonstrates the size and function of various chambers of the heart.
* The stress test involves exercise using a treadmill or a stationary bike. In patients who are unable to complete a high level of exercise due to physical limitations, stress to the heart is provided by a pharmaceutical or chemical stimulation to the heart. Exercise is started at a slower, warm-up speed and then increased every 3 minutes. Exercise is abruptly stopped once the patient exceeds 85% of the target rate. EKG recordings are made every minute of exercise and then again after exercise is stopped. Blood pressure is recorded at three minute intervals during exercise and then again at rest.
* Immediately after exercise is stopped, the patient will undergo a repeat echocardiogram.
* If no cardiac abnormalities are detected, the screening tests will be repeated every 3 years, if the patient is less than 10 years out from their initial treatment. If the patient is more than 10 years from initial treatment, then the tests will be repeated at approximately 18 months from the initial screening and once more at the end of the third year.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at Brigham and Women's Hospital or Dana-Farber Cancer Institute for Hodgkin's disease with mediastinal irradiation
* Age > or = to 15 years of age
* Five years or longer after initial treatment
* Relapse-free interval of > 1 year

Exclusion criteria:

* Patients treated for Hodgkin's disease outside of Brigham and Women's Hospital or Dana-Farber Cancer Institute
* Current age < 15 years of age
* Less than 5 years out from initial treatment
* Relapses within 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2004-02; Primary Completion 2007-10 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of a cardiac screening program in patients who are 5 to 10 years our from initial mediastinal irradiation for Hodgkin's disease. | 3 years
  Compliance of screening and follow up visits are tracked

SECONDARY OUTCOMES:
To prospectively collect data on the prevalence of modifiable cardiac risk factors and the spectrum of cardiac structural abnormalities in this patient populations | 3 years
  Data on modifiable cardiac risk factors, and outcome of screening studies, are collected prospectively
to correlate cardiac structural abnormalities with quality of life | 3 years
  Responses to the generic quality-of-life questionnaire Short-Form 36 (SF-36) collected at the time of initial visit, will be correlated with cardiac screening results
to correlate cardiac structural abnormalities with level of fatigue. | 3 years
  Responses to the fatigue subscale of FACT-Fatigue (FACT-F), collected at the time of initial visit, will be correlated with cardiac screening results

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K. Ng, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No